CLINICAL TRIAL: NCT05343624
Title: Use of Continuous Glucose Monitors in Coronavirus Disease 2019 ICU and Potential Inpatient Settings
Acronym: CGMCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20200558
Record Dates: First submitted 2021-08-03; First posted 2022-04-25 (Actual); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Covid19; Diabetes Mellitus
MeSH Terms: conditions — COVID-19; Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CGM Arm (Other): continuous glucose meter is placed on the abdomen
  Interventions: Device: continuous glucose monitoring

INTERVENTIONS:
Device: continuous glucose monitoring — Use of continuous glucose monitoring in inpatient and ICU settings

SUMMARY:
The objective of the study is to improve glycemic control in inpatient/ICU settings using real- time continuous glucose monitors (CGM) data for insulin titration. It may help reduce Coronavirus disease 2019 patient contact with healthcare workers as well.

DETAILED DESCRIPTION:
Due to the increasing need for acute care of COVID-19 patients in ICU settings, the use of continuous glucose monitors (CGM) as a means to reduce patient contact and remotely improve glycemic control for diabetic COVID-19 patients needs to be explored. As demonstrated by recent data published in China, Wuhan province patients with diabetes made up 22.2% of COVID-19 ICU patient populations with a subsequent mortality of 7.3% (3). Not only during COVID-19 pandemic but also previous experiences with SARS and influenza viral respiratory infections demonstrated increased mortality in those patients with hyperglycemia (4).

Using CGMs provides timely access to glucose trends, commonly used to determine insulin dosing decisions in outpatient settings (5). Implementing their use for hospitalized patients could be expected to improve healthcare worker insight into glycemic control therapies.

Considering the ease of transmission of the SARS-Cov-2 virus, it is important to minimize duration and frequency of patient contact in order to maintain the safety of COVID-19 healthcare workers without compromising on their glycemic control. The WHO recommends that any healthcare provider coming into direct contact with COVID-19 patients should be utilizing appropriate PPE for each encounter. In this time of limited PPE supply (6), remote glucose monitoring can allow for rational use of these limited resources. With appropriate training on CGM data interpretation, nursing and ordering providers could expect to develop and implement more efficient insulin plans, requiring fewer physical contact with COVID-19 positive patients.

ELIGIBILITY:
Inclusion Criteria:

* Coronavirus disease 2019 tested positive patient
* Age over 18 years
* Admitted to Coronavirus disease 2019 specific ICU, with possible transfer to inpatient unit when stable
* Patients with known or acquired Type 1 or Type 2 Diabetes requiring insulin therapy during admission

Exclusion Criteria:

* In state of active diabetic ketoacidosis (DKA) at time of enrollment
* Two or more vasopressors in use at time of sensor placement
* Unable to use at predetermined sensor site based on assessment of skin health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CGM Arm
Started | 9
Completed | 8
Not Completed | 1
Not completed — Chart review not completed | 1

BASELINE CHARACTERISTICS:
Population: No data was collected on race or ethnicity.
Arm/Group | CGM Arm
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time in Range
Description: Percentage of time spent in target glucose range of 140-180mg/dL
Time Frame: 14 days
Measure: Median (Standard Deviation); unit: percentage of time
Arm/Group | CGM Arm
Number analyzed (Participants) | 8
percentage of time | 21.6 (13.47)

2. Secondary Outcome: Number of Days CGM Worn
Description: Number of days the CGM was worn
Time Frame: 14 days
Measure: Median (Standard Deviation); unit: days
Arm/Group | CGM Arm
Number analyzed (Participants) | 8
days | 5 (5.39)

3. Secondary Outcome: Hypoglycemia
Description: Average number of hypoglycemia events per participant
Time Frame: 14 days
Measure: Median (Standard Deviation); unit: Events
Arm/Group | CGM Arm
Number analyzed (Participants) | 8
Events
  Low 54-140mg/dl | 13.8 (10.44)
  Very low <54 mg/dl | 0 (1.07)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | CGM Arm
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT05343624/Prot_SAP_001.pdf